CLINICAL TRIAL: NCT02185313
Title: Verticality Perception and Gaze Holding in Healthy Human Subjects and Patients With Acute and Chronic Cerebellar Disorders
Brief Title: Gaze Holding in Cerebellar Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: gaze_holding_cerebellar_zurich
Record Dates: First submitted 2014-07-02; First posted 2014-07-09 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Gaze Holding in Humans; Rebound in Humans

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gaze holding (Experimental)
  Interventions: Other: visual stimulus to follow

INTERVENTIONS:
Other: visual stimulus to follow

SUMMARY:
The long-term goal of this research is to advance the investigators knowledge of how the cerebellum a) controls gaze holding and compensates for impaired gaze stability and b) modulates vestibular information that is forward-ed from the labyrinth and brought to perception. While gaze holding is stable also at large angles of gaze eccentricity in healthy human subjects, patients with chronic (degenerative) cerebellar disorders are inable to stabilize gaze in eccentric positions, resulting in eye drift towards primary (straight-ahead) position and com-pensatory gaze-evoked nystagmus. When returning to primary position, a compensatory nystagmus into the opposite direction (called rebound nystagmus) can be observed in these patients. Unlike patients with de-generative cerebellar disorders, patients suffering from ischemic of hemorrhagic stroke within the cerebellum present with acute deficits of gaze holding and verticality perception.

While a linear relationship between the amount of eye velocity drift and eccentricity of eye position has been proposed in healthy human subjects, others suggested non-linear behaviour. The strategy of this research is to characterize gaze holding and verticality perception in healthy human subjects and patients with either acute (ischemic or hemorrhagic) or chronic degenerative cerebellar disorders and to relate eye movement findings with structural imaging of the cerebellum. The investigators will therefore analyze key cerebellar structures with regards to loss of volume and relate these imaging findings with the participants' ability to hold gaze and es-timate direction of vertical. The investigators hypothesize that besides the flocculus other vestibulo-cerebellar structures are involved in gaze holding and verticality perception in humans.

ELIGIBILITY:
Inclusion Criteria:

1. ages 18-85
2. informed consent
3. for group 1: acute (i.e. symptom onset <14 days ago) cerebellar ischemia or hemorrhage as confirmed by clinical examination and brain imaging (CT or MRI)
4. for group 2: chronic cerebellar degeneration as confirmed by clinical examination (presence of downbeat-nystagmus and / or gaze-evoked nystagmus and / or ataxia of gait and stance) in the absence of focal lesions (as previous cerebellar stroke, mass lesion or inflammation) on clinical routine cerebellar imaging
5. absence of exclusion criteria

Exclusion Criteria:

1. has MRI contraindications such as pacemaker, implanted pumps, shrapnel, etc. (full MRI screening form will be filled out).
2. disturbed consciousness
3. other neurological or systemic disorder which can cause dementia or cognitive dysfunction
4. Pregnancy or possible pregnancy if not ruled out by a negative pregnancy test.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
eye velocity in relation to eye position | during the visual stimulus (5min)

SECONDARY OUTCOMES:
symmetry of eye velocity for right vs. left gaze | during the visual stimulus (5min)

CONTACTS AND LOCATIONS:
Overall Officials: Dominik Straumann, Prof MD, Principal Investigator — University Hospital Zurich, Division of Neurology
Locations (1):
- University Hospital Zurich, Division of Neurology, Zurich, Canton of Zurich, Switzerland